CLINICAL TRIAL: NCT03488199
Title: Independent Randomized Trial in Carotid Artery Revascularization Comparing the Stent (Acculink™) Versus the Mesh Covered Stent (CGuard™) The SIBERIA Trial
Brief Title: The SIBERIA Trial (Acculink™ Versus CGuard™)
Acronym: CAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRICP 9872
Record Dates: First submitted 2017-09-12; First posted 2018-04-04 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-09

CONDITIONS: Patients With Aterosclerotic Carotid Stenosis; Symptomatic Patients (Stenosis > 50%); Asymptomatic Patients (Stenosis ≥80%)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stent Acculink™ (RX ACCULINK CAROTID STENT SYSTEM) (Active Comparator): 50 Carotid stenting (RX ACCULINK CAROTID STENT SYSTEM)
  Interventions: Device: Stent Acculink ™
- Stent CGuard™ (The CGuardTM Embolic Prevention System (EPS)) (Experimental): 50 Carotid stenting (The CGuardTM Embolic Prevention System (EPS))
  Interventions: Device: CGuardTM™

INTERVENTIONS:
Device: Stent Acculink ™ — Carotid Artery Revascularization using Stents
  Other Names: RX ACCULINK CAROTID STENT SYSTEM
  Arms: Stent Acculink™ (RX ACCULINK CAROTID STENT SYSTEM)
Device: CGuardTM™ — Carotid Artery Revascularization using Stents
  Other Names: The CGuardTM Embolic Prevention System (EPS)
  Arms: Stent CGuard™ (The CGuardTM Embolic Prevention System (EPS))

SUMMARY:
That the study will be carried out as it has the protocol instructions, respecting the applicable regulations for clinical investigations with medical devices and following the internationally accepted ethical standards

DETAILED DESCRIPTION:
Independent Randomized Trial in Carotid Artery Revascularization Comparing the Stent (Acculink™) Versus the Mesh Covered Stent (CGuard™) was performed.

Ischemic lesions of brain after CAS were determined by MRI before and after treatment (2-3 days, 1 month).

ELIGIBILITY:
Inclusion Criteria

1. Consecutive patients 45-80 years old accepted for CAS following neurological consultation and qualification for the procedure according to center's routine practice.
2. More than 6-month life expectancy
3. Suitable clinical conditions for performing DW-MRI
4. Written Informed consent approved by the Ethics Committee
5. Subject agrees to all required follow-up procedures and visits

Exclusion Criteria:

1. Currently enrolled in another investigational device or drug study that has not completed the study or that clinically interferes with the current study endpoints
2. Recent surgical procedure within 30-days before or planned surgery within 30-days after the stenting procedure
3. Hepatic active disease (bilirubin> 35 mmol / l) or renal insufficiency (serum creatinine > 2.5 mg/dL or glomerular filtration rate <60 ml / min)
4. Recent evolving acute stroke within 30-days of study evaluation
5. Myocardial infarction within 72 hours prior to carotid stenting procedure (CPK-MB > 3 times normal)
6. Female patients of childbearing potential or known to be pregnant
7. Any known factor for potential stroke other than carotid stenosis, such as atrial fibrillation or atrial flutter (paroxysmal, permanent or persistent) or thrombophilia
8. Patient on VKA or new oral anticoagulants

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-03-09 (Actual)

PRIMARY OUTCOMES:
determination of ischemic lesions | at 30-days
  New DW-MRI lesions post procedural their permanence at 30-days
determination of ischemic lesions | at 48 hours
  New DW-MRI lesions post procedural (48 hours)

CONTACTS AND LOCATIONS:
Locations (1):
- Andrey A. Karpenko, Novosibirsk, Russia

REFERENCES:
- [Derived] Karpenko A, Bugurov S, Ignatenko P, Starodubtsev V, Popova I, Malinowski K, Musialek P. Randomized Controlled Trial of Conventional Versus MicroNet-Covered Stent in Carotid Artery Revascularization. JACC Cardiovasc Interv. 2021 Nov 8;14(21):2377-2387. doi: 10.1016/j.jcin.2021.08.005. PMID 34736737